CLINICAL TRIAL: NCT01902420
Title: Investigation of Prevalence and Clinical Effects of Aryl Hydrocarbon Receptor Interacting Protein (AIP) Gene Mutations With DNA Sequence Analysis in Acromegaly Patients in Turkey
Brief Title: Aryl Hydrocarbon Receptor Interacting Protein (AIP) Gene Mutations in Acromegaly
Acronym: AIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ZULEYHA KARACA, Assoc. Prof Dr Zuleyha KARACA, TC Erciyes University
Other Study IDs: 113S432
Record Dates: First submitted 2013-07-12; First posted 2013-07-18 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with acromegaly: patients with acromegaly caused by a growth hormone secreting pituitary adenoma
- healthy control: healthy volunteers without a personal or family history of pituitary adenoma

SUMMARY:
Acromegaly is a rare disease caused by growth hormone (GH) secreting pituitary adenoma in more than 95% of cases. Acromegaly can be seen sporadically or may be associated with a variety of genetic syndromes such as Multiple Endocrine Neoplasia Type 1, Carney Complex, familial isolated pituitary adenoma (FIPA) and Mc-Cune Albright Syndrome. The accompanying features of these syndromes and family history are helpful in the differential diagnosis. Aryl hydrocarbon receptor (AHR)-interacting protein (AIP) gene mutations can be seen sporadically as well as in FIPA. But the prescience of the presence of AIP mutation is limited by positive family history and early-onset of acromegaly. Furthermore, the probability of the patient to be the index case of the family should not be ignored.

Screening for AIP gene mutation is recommended in patients with pituitary adenomas of childhood-onset, GH or prolactin secreting tumors who are diagnosed before the age of 30 years and positive family history in two or more family members according to present evidence in the literature. It is also known that AIP mutation is usually associated with more aggressive clinical behavior due to unclarified reasons.

The prevalence of AIP mutation in Turkish population and types of mutations have not been defined previously. The primary aim of the present study is to define the AIP gene mutation prevalence and the relation with clinical and tumour behaviour in a subgroup of Turkish acromegalic patients. If AIP gene mutation is detected in some patients, it will be possible to screen the family of the patient for the presence of AIP mutation or at least for the presence of pituitary adenoma.

Acromegalic patients who are followed in Erciyes University Medical School Department of Endocrinology will be enrolled into the study. After DNA isolation, each exon of AIP gene including splicing points will be reproduced by polymerase chain reaction (PCR) and will be analyzed for the presence of mutation by sequence analysis. The cases will be analyzed further in means of clinical features according to presence of AIP gene mutation.

The prevalence of AIP gene mutation, clinical reflection of presence of AIP mutation will be determined and genetic consultation will be given to the carriers of AIP gene mutation at the end of the study.

DETAILED DESCRIPTION:
Screening for AIP gene mutation is recommended in patients with pituitary adenomas of childhood-onset, GH or PRL secreting tumors who are diagnosed before the age of 30 years and positive family history in two or more family members according to present evidence in the literature. It is also known that AIP mutation is usually associated with more aggressive clinical behavior due to unclarified reasons.

The prevalence of AIP mutation in Turkish population and types of mutations have not been defined previously. The primary aim of the present study is to define the AIP gene mutation prevalence and the relation with clinical and tumour behavior in a subgroup of Turkish acromegalic patients. If AIP gene mutation is detected in some patients, it will be possible to screen the family of the patient for the presence of AIP mutation or at least for the presence of pituitary adenoma.

Acromegalic patients who are followed in Erciyes University Medical School Department of Endocrinology will be enrolled into the study. The clinical and laboratory data will be recorded and the remission status of the patients will be determined. Each exon of AIP gene including splicing points will be reproduced by PCR and will be analyzed for the presence of mutation by sequence analysis. Genomic DNA will be isolated from peripheral blood samples of acromegalic patients by using the QIAamp DNA blood mini kit (QIA-GEN, Milano, Italy) according to the manufacturer's instruction. Fifty nanograms of genomic DNA will be ampliﬁed with primers as reported. The entire AIP gene will be examined acromegaly patients and healthy control group. Each AIP exon from each DNA sample will be ampliﬁed using PCR. Six AIP exons will be ampliﬁed using the Thermo Taq DNA polymerase and following conditions: an initial denaturation at 96°C for 5 min, followed by 34 cycles of 94°C for 45 s, 60°C for 45 s, 72°C for 1 min, then a ﬁnal extension step at 72°C for 7 min.PCR ampliﬁcations will be checked on a 2 % agarose gel. PCR products will be purified by PCR purification kit. Sequential alterations will be determined by bidirectional sequencing. Six AIP exons will be sequenced by using Beckman CEQ 8000.

The cases will be analyzed further in means of clinical features according to presence of AIP gene mutation.

The prevalence of AIP gene mutation, clinical reflection of presence of AIP mutation will be determined and genetic consultation will be given to the carriers of AIP gene mutation at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acromegaly

Exclusion Criteria:

* Patients with acromegaly due to ectopic GH or GHRH secreting tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: acromegaly patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
number of acromegalic patients with AIP mutation | up to 18 months

SECONDARY OUTCOMES:
number of acromegalic patients with aggressive tumor with AIP mutation | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Zuleyha Karaca, Principal Investigator — Erciyes University Medical School Department of Endocrinology Kayseri/Turkey; Serpil Taheri, Principal Investigator — Erciyes University Medical School Department of Medical Biology, Kayseri/Turkey; Fahrettin Kelestimur, Study Director — Erciyes University Medical School Department of Endocrinology Kayseri/Turkey; Fatih Tanriverdi, Study Chair — Erciyes University Medical School Department of Endocrinology Kayseri/Turkey; Kursad Unluhizarci, Study Chair — Erciyes University Medical School Department of Endocrinology Kayseri/Turkey
Locations (1):
- Erciyes University Medical School Department of Endocrinology, Kayseri, Turkey (Türkiye)